CLINICAL TRIAL: NCT03837522
Title: Pilot Randomized Trial to Define the Benefits and Harms of Deceased Donor Kidney Procurement Biopsies
Brief Title: Trial to Define the Benefits and Harms of Deceased Donor Kidney Procurement Biopsies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: Mid-America Transplant (Other); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Krista Lentine MD, PhD, Professor, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 29880
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Kidney Transplant; Renal Transplant
Keywords: Biopsy; Deceased kidney donation; Kidney transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Procurement Biopsy: Frozen section (Active Comparator): In the routine care condition, biopsies will be processed immediately as a frozen section.
  Interventions: Diagnostic Test: Procurement Biopsy: Frozen section
- Procurement Biopsy: Permanent section (Active Comparator): In the intervention group, the biopsy processing will be delayed to permanent section, and therefore not available until allocation is complete.
  Interventions: Diagnostic Test: Procurement Biopsy: Permanent section

INTERVENTIONS:
Diagnostic Test: Procurement Biopsy: Frozen section — Frozen sections are prepared by freezing and slicing the tissue sample; importantly, they can be done in about 15 to 20 minutes. Frozen sections are done when an immediate answer is needed, but do not provide optimal quality.
  Other Names: Immediate results
  Arms: Procurement Biopsy: Frozen section
Diagnostic Test: Procurement Biopsy: Permanent section — Permanent sections are prepared by placing the tissue in fixative (usually formalin) to preserve the tissue, processing it through additional solutions, and then placing it in paraffin wax. After the wax has hardened, the tissue is cut into very thin slices, which are placed on slides and stained. The process normally takes several days.
  Other Names: Delayed results
  Arms: Procurement Biopsy: Permanent section

SUMMARY:
The purpose of this research study is to compare the impact of the availability of biopsy results at the time of organ offers on the use and outcomes of kidneys from deceased donors.

DETAILED DESCRIPTION:
Randomization of biopsy processing will be performed at the level of the deceased donor.

If the participant agrees to be in this study and signs the informed consent, at the time that a kidney is accepted for them, the accepted deceased donor will be randomized, like a flip of a coin, to one of two groups.

* Group 1: biopsies will be processed immediately (routine "frozen section") and results will be available to clinical teams at the time of the organ offers. Frozen section refers to a process where tissue from the biopsy sample is prepared by freezing and then slicing the tissue sample. Importantly, it can be done in about 15 to 20 minutes. Frozen sections are done when an immediate answer is needed; however, the quality of the sample is not always optimal.
* Group 2: biopsies will be processed using "permanent sections" - these results will not be available until after the organ is transplanted. Permanent section refers to a process where tissue from the biopsy sample is prepared by placing the tissue sample in a fixative, called formalin, to preserve the tissue, processing it through other additional solutions, and then placing it in paraffin wax. After the wax hardens, the tissue is cut into very thin slices, which are placed on slides and stained. This process normally takes several days.

There is a 50/50 chance that the donor will be randomized to immediate biopsy processing by frozen section, versus permanent processing that yields results after transplant. If for any reason their surgeon feels that it would not be safe to proceed without the biopsy result, he or she will have the ability to receive the results of the biopsy before the transplant. The study team will record any episodes of this occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant candidate
* On waitlist for kidney transplant at the time of informed consent at one of the participating sites
* Age 18 or older
* Willing and able to provide informed consent for participation in the study

Exclusion Criteria:

* Unable or unwilling to provide informed consent to participate in the study
* Younger than 18 years old
* Not on waitlist for kidney transplant at the time of informed consent at one of the participating centers
* Candidates for or recipients of multi-organ transplants (kidney along with another solid organ)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-02-04 (Actual)

PRIMARY OUTCOMES:
risk-adjusted kidney yield | 3 years
  per kidney donor with an immediate vs delayed procurement biopsy processing (this will serve as the primary organ utilization metric, and is the adjusted converse of organ discard)

SECONDARY OUTCOMES:
Life years for transplant recipients | 3 years
  Life years or survival for candidates after offer of kidney with an immediate vs delayed procurement biopsy processing
Number of participants with delayed graft function | 3 years
  Number of participants with delayed graft function after transplant of kidney with an immediate vs delayed procurement biopsy processing
Number of participants with graft survival | 3 years
  Number of participants with graft survival after transplant of kidney with an immediate vs delayed procurement biopsy processing
Cold ischemia time | 3 years
  Cold ischemia time for kidneys transplanted after immediate vs delayed procurement biopsy processing
Patient survival after transplant | 3 years
  Patient survival after transplant of kidney with an immediate vs delayed procurement biopsy processing

CONTACTS AND LOCATIONS:
Overall Officials: Krista Lentine, MD, PhD, Principal Investigator — St. Louis University
Locations (2):
- United States (2):
  - Saint Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri

REFERENCES:
- [Background] Cooper M, Formica R, Friedewald J, Hirose R, O'Connor K, Mohan S, Schold J, Axelrod D, Pastan S. Report of National Kidney Foundation Consensus Conference to Decrease Kidney Discards. Clin Transplant. 2019 Jan;33(1):e13419. doi: 10.1111/ctr.13419. Epub 2018 Oct 21. PMID 30345720
- [Background] Wang CJ, Wetmore JB, Crary GS, Kasiske BL. The Donor Kidney Biopsy and Its Implications in Predicting Graft Outcomes: A Systematic Review. Am J Transplant. 2015 Jul;15(7):1903-14. doi: 10.1111/ajt.13213. Epub 2015 Mar 13. PMID 25772854
- [Background] Naesens M. Zero-Time Renal Transplant Biopsies: A Comprehensive Review. Transplantation. 2016 Jul;100(7):1425-39. doi: 10.1097/TP.0000000000001018. PMID 26599490
- [Background] Hart A, Smith JM, Skeans MA, Gustafson SK, Stewart DE, Cherikh WS, Wainright JL, Kucheryavaya A, Woodbury M, Snyder JJ, Kasiske BL, Israni AK. OPTN/SRTR 2015 Annual Data Report: Kidney. Am J Transplant. 2017 Jan;17 Suppl 1(Suppl 1):21-116. doi: 10.1111/ajt.14124. PMID 28052609
- [Background] De Vusser K, Lerut E, Kuypers D, Vanrenterghem Y, Jochmans I, Monbaliu D, Pirenne J, Naesens M. The predictive value of kidney allograft baseline biopsies for long-term graft survival. J Am Soc Nephrol. 2013 Nov;24(11):1913-23. doi: 10.1681/ASN.2012111081. Epub 2013 Aug 15. PMID 23949799
- [Background] Kasiske BL, Stewart DE, Bista BR, Salkowski N, Snyder JJ, Israni AK, Crary GS, Rosendale JD, Matas AJ, Delmonico FL. The role of procurement biopsies in acceptance decisions for kidneys retrieved for transplant. Clin J Am Soc Nephrol. 2014 Mar;9(3):562-71. doi: 10.2215/CJN.07610713. Epub 2014 Feb 20. PMID 24558053
- [Background] Husain SA, Chiles MC, Lee S, Pastan SO, Patzer RE, Tanriover B, Ratner LE, Mohan S. Characteristics and Performance of Unilateral Kidney Transplants from Deceased Donors. Clin J Am Soc Nephrol. 2018 Jan 6;13(1):118-127. doi: 10.2215/CJN.06550617. Epub 2017 Dec 7. PMID 29217537
- [Background] Hart A, Smith JM, Skeans MA, Gustafson SK, Wilk AR, Robinson A, Wainright JL, Haynes CR, Snyder JJ, Kasiske BL, Israni AK. OPTN/SRTR 2016 Annual Data Report: Kidney. Am J Transplant. 2018 Jan;18 Suppl 1(Suppl 1):18-113. doi: 10.1111/ajt.14557. PMID 29292608
- [Background] Walker PD, Cavallo T, Bonsib SM; Ad Hoc Committee on Renal Biopsy Guidelines of the Renal Pathology Society. Practice guidelines for the renal biopsy. Mod Pathol. 2004 Dec;17(12):1555-63. doi: 10.1038/modpathol.3800239. PMID 15272280
- [Derived] Lentine KL, Kasiske B, Axelrod DA. Procurement Biopsies in Kidney Transplantation: More Information May Not Lead to Better Decisions. J Am Soc Nephrol. 2021 Aug;32(8):1835-1837. doi: 10.1681/ASN.2021030403. Epub 2021 May 27. No abstract available. PMID 34045315
- See also: National Kidney Foundation. Progress: Discarding a kidney can discard a life. Overview of Consensus Conference to Decrease Kidney Discards. — https://www.kidney.org/newsletter/board-to-board/progress-discarding-kidney-can-discard-life
- See also: Eurotransplant Statistics Report Library. — http://statistics.eurotransplant.org